CLINICAL TRIAL: NCT01858623
Title: Pharmacokinetic Interactions of Losartan and Hydrochlorothiazide
Acronym: PKLH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damanhour University (Other)
Responsible Party: Principal Investigator, Sally Helmy, PhD, CPHQ, Lecturer of Pharmaceutics, Faculty of Pharmacy, Damanhour University
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: PPT5
Record Dates: First submitted 2013-05-12; First posted 2013-05-21 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: Healthy Normotensive Participants
Keywords: Healthy Normotensive Participants; Fixed dose combination; Pharmacokinetics; Losartan; Hydrochlorothiazide
MeSH Terms: interventions — hydrochlorothiazide, losartan drug combination; Losartan; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Losartan / Hydrochlorothiazide100 mg/25mg (Other): Losartan / Hydrochlorothiazide100 mg/25mg fixed dose combination
  Interventions: Drug: Losartan/hydrochlorothiazide
- Losartan 100 mg (Other): Losartan 100 mg alone
  Interventions: Drug: Losartan
- hydrochlorothiazide 25 mg (Other): hydrochlorothiazide 25 mg alone
  Interventions: Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Losartan/hydrochlorothiazide
  Arms: Losartan / Hydrochlorothiazide100 mg/25mg
Drug: Losartan
  Arms: Losartan 100 mg
Drug: Hydrochlorothiazide
  Arms: hydrochlorothiazide 25 mg

SUMMARY:
This study was conducted to investigate any potential reaction between losartan and hydrochlorothiazide.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old and not more than 45 healthy male volunteers
* Who had passed all the screening parameters

Exclusion Criteria:

* A clinically significant abnormal physical exam, medical history, or laboratory studies
* If they showed a sitting SBP of >140 or <100 mmHg, DBP > 90 or <60mm Hg, or a pulse rate of > 95 or < 50 beats/min at screening
* The use of any prescription drug within the previous month or use of any over-the-counter medication within the past 14 days
* A history of blood dyscrasias
* A history of alcohol or drug abuse within the past year
* Donation of blood during the 8 weeks prior to the study or plans to donate blood during or within 8 weeks of completing the study
* Unable to tolerate vein puncture and multiple blood samplings
* Any surgical/medical condition that might alter drug absorption, distribution, metabolism, or excretion

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2013-02; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Heart rate | Participants will be followed for the duration of study, an expected average of 5 weeks.
Blood pressure | Participants will be monitored for the duration of study, an expected average of 5 weeks.
Pharmacokinetic parameter such as Cmax of losartan and hydrochlorothiazide | At the end of the study, after collection of all blood samples, an expected average of 4 weeks
Pharmacokinetic parameter such as AUC of losartan and hydrochlorothiazide | At the end of the study, after collection of all blood samples, an expected average of 4 weeks